CLINICAL TRIAL: NCT01598077
Title: A Phase I Study of LJM716 in Patients With Squamous Cell Carcinoma of Head and Neck, or HER2 Overexpressing Metastatic Breast Cancer or Gastric Cancer
Brief Title: A Phase I Study of LJM716 in Squamous Cell Carcinoma of Head and Neck, or HER2+ Breast Cancer or Gastric Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLJM716X2101; 2011-004865-33 (EudraCT Number)
Record Dates: First submitted 2012-05-04; First posted 2012-05-15 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2014-04

CONDITIONS: HER2 + Breast Cancer, HER2 + Gastric Cancer, Squamous Cell Carcinoma of Head and Neck, Esophageal Squamous Cell Carcinoma; HER2 + Breast Cancer; HER2 + Gastric Cancer; Squamous Cell Carcinoma of Head and Neck; Esophageal Squamous Cell Carcinoma
Keywords: Breast cancer, gastric cancer, squamous cell carcinoma of head and neck, esophageal squamous cell carcinoma; Breast cancer; Gastric cancer; Squamous cell carcinoma of head and neck; Esophageal squamous cell carcinoma
MeSH Terms: conditions — Breast Neoplasms; Stomach Neoplasms; Esophageal Squamous Cell Carcinoma; Squamous Cell Carcinoma of Head and Neck | interventions — elgemtumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dose escalation and dose expansion (Experimental)
  Interventions: Drug: LJM716

INTERVENTIONS:
Drug: LJM716

SUMMARY:
This primary purpose of this study is to estimate the maximum tolerated dose (MTD) and/or recommended dose for expansion (RDE) and preferred dosing schedule of LJM716 given by IV infusion in adult patients with squamous cell carcinoma of head and neck, or esophagus, or HER2 overexpressing metastatic breast cancer or gastric cancer

ELIGIBILITY:
Inclusion criteria:

* Patients with HER2+ breast cancer, or HER2+ gastric cancer, or squamous cell carcinoma of head and neck, or esophageal squamous cell carcinoma
* Site of disease that can be safely biopsied

Exclusion criteria:

* Patients received prior anti-HER3 antibody treatment
* Patients with impaired cardiac function
* Brain metastases that have not been adequately treated
* Malignant disease other than that being treated in this study
* Pregnant or nursing (lactating) women
* Laboratory abnormalities as specified in the protocol Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2012-07; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLTs) | 4 weeks

SECONDARY OUTCOMES:
Adverse events | 4 months
Serious adverse events | 4 months
Pharmacodynamic response to LJM716 in tumor tissue | 3 months
Frequency of partial responses, complete responses and stable disease according to RECIST | every 2 months
Serum concentration of antibodies to LJM716 | 18 months
Progression-free survival | 18 months
Duration of response | 18 months
Serum concentration of LJM716, | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (8):
- United States (4):
  - University of Chicago Medical Center University of Chicago (16), Chicago, Illinois
  - Massachusetts General Hospital SC-5, Boston, Massachusetts
  - University of Texas/MD Anderson Cancer Center UT MD, Houston, Texas
  - University of Utah / Huntsman Cancer Institute Huntsman, Salt Lake City, Utah
- Novartis Investigative Site, Toronto, Ontario, Canada
- Novartis Investigative Site, Seoul, Korea, South Korea
- Novartis Investigative Site, Barcelona, Catalonia, Spain
- Novartis Investigative Site, Taipei, Taiwan

REFERENCES:
- [Derived] Reynolds KL, Bedard PL, Lee SH, Lin CC, Tabernero J, Alsina M, Cohen E, Baselga J, Blumenschein G Jr, Graham DM, Garrido-Laguna I, Juric D, Sharma S, Salgia R, Seroutou A, Tian X, Fernandez R, Morozov A, Sheng Q, Ramkumar T, Zubel A, Bang YJ. A phase I open-label dose-escalation study of the anti-HER3 monoclonal antibody LJM716 in patients with advanced squamous cell carcinoma of the esophagus or head and neck and HER2-overexpressing breast or gastric cancer. BMC Cancer. 2017 Sep 12;17(1):646. doi: 10.1186/s12885-017-3641-6. PMID 28899363
- See also: Results for CLJM716X2101 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=13604